CLINICAL TRIAL: NCT03132376
Title: Effects of Consuming Protein Shakes, Varying in Protein Source, on Appetite, Satiety and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MU2005830
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breakfast Preload Drink (Experimental): Participants were given isovolumetric drinks, to consume in the morning after an overnight fast, followed by questionnaires asking throughout the day asking participants of their perceived hunger, fullness, desire to eat, and prospective food consumption, and if they would like to eat again. Four hours following consumption, they were given an ad libitum pasta meal to consume.
  The drinks consisted of the following:
  Water Preload Drink, Whey Protein Isolate Drink, Micellar Casein Protein Drink, Egg White Isolate Protein Drink, and Egg White Concentrate Protein Drink
  Interventions: Dietary Supplement: Water Preload Drink; Dietary Supplement: Whey Protein Isolate Drink; Dietary Supplement: Micellar Casein Protein Drink; Dietary Supplement: Egg White Isolate Protein Drink; Dietary Supplement: Egg White Concentrate Protein Drink

INTERVENTIONS:
Dietary Supplement: Water Preload Drink — Participants were given 275 ml (0 kcal) water to consume in the morning following an overnight fast. This served as the control drink.
Dietary Supplement: Whey Protein Isolate Drink — Participants were given an isovolumetric (to the water), 160 kcal drink with 30 g whey protein to consume in the morning following an overnight fast.
Dietary Supplement: Micellar Casein Protein Drink — Participants were given an isovolumetric (to the water), 160 kcal drink with 30 g micellar casein to consume in the morning following an overnight fast.
Dietary Supplement: Egg White Isolate Protein Drink — Participants were given an isovolumetric (to the water), 160 kcal drink with 30 g egg white isolate protein to consume in the morning following an overnight fast.
Dietary Supplement: Egg White Concentrate Protein Drink — Participants were given an isovolumetric (to the water), 160 kcal drink with 30 g egg white concentrate protein to consume in the morning following an overnight fast.

SUMMARY:
Background: Consistent data from acute, single preload studies demonstrate improvements in perceived appetite and satiety following the consumption of high-protein preloads compared to normal protein preloads. However, it is currently unclear as to whether protein quality (i.e., protein source) or the use of appetite questionnaires influences these outcomes. Objective: To examine whether the consumption of protein preloads (egg white isolate, whey isolate, micellar casein, and instant egg white) differentially modulate postprandial hunger, fullness, desire to eat, prospective food consumption, eating initiation, and subsequent food intake; and if the use of appetite questionnaires to assess perceived appetite and satiety affect subsequent energy intake. Methods: Twelve young adults (age: 22±1 y; BMI: 22.1±0.9 kg/m2) reported to the research facility between 7 - 9 am to complete each 4-h testing day. A set of questionnaires assessing perceived hunger, fullness, desire to eat, prospective food consumption were completed followed by the consumption of the 130 kcal beverage preloads, varying in protein source. A water preload was also included as a control. The same set of questionnaires along with the assessment of whether they would like to eat again were completed every 30 min throughout the 4-h postprandial period. On a separate day, all twelve young adults also completed a similar testing day except were not given questionnaires throughout the 4-h postprandial period. After the 4-h, the participants were given an ad libitum pasta meal to consume until 'comfortably full.' Results: The consumption of the protein preloads improved hunger, fullness, desire to eat, prospective food consumption and delayed the request to eat again vs. the control (water); however, no differences in appetite and satiety outcomes were observed between protein sources. No differences in energy content at the lunch meal were observed between any preloads. The use of questionnaires did not change energy consumed at the lunch meal. Conclusions: When comparing high-quality animal-based proteins consumed as a beverage preload, relatively no differences in markers of appetite control and satiety were detected, suggesting that protein quality has little impact on these outcomes when consuming 30g of protein. In addition, the use of questionnaires assessing perceived appetite and satiety do not impact subsequent energy intake.

DETAILED DESCRIPTION:
the following acute, randomized crossover study will be completed in 12 healthy adults (age 18-35y; BMI: 18-29.9 kg/m2) to compare 135 kcal protein beverages consumed at breakfast containing 30 g of protein from whey isolate (WY), casein (CS), egg white isolate (EWI), egg white protein concentrate (EWP), or a 0 kcal water beverage - which serves as the control (CON). Note: the W beverage will be consumed on 2 different days; these days only differ by the postprandial outcomes completed (see below).

The participants will report to the research facility between 7 - 9 am to complete each 4-h testing day. Prior to testing, the participants will be provided with a standardized dinner to consume, at home, between 5-7 pm the night before each testing day. Upon arrival to the facility, each participant will become familiarized with the testing day procedures. At time -15 min, a baseline set of computerized questionnaires will be completed. At time 0 min, one of the breakfast beverages will be provided. Immediately following the first swallow of the breakfast shakes, the participants will be given a questionnaire assessing the palatability of each shake. The participants will consume the beverage within 20 min. For 5 of the 6 days, a set of questionnaires will be completed every 30 min throughout the 4-h postprandial period. For one of the W days, no questionnaires will be completed. After the 4-h, the participants will be given an ad libitum pasta meal to assess energy intake. For the lunch meal, the participants will be given 30 min to "consume as much or as little as possible until comfortably full." Following these procedures, the participants will be allowed to leave the facility. The next day, a dietary recall will be performed to assess daily energy intake following the consumption of the previous day's breakfast beverage.

ELIGIBILITY:
Inclusion Criteria:

1. healthy
2. ages 18-35 years old
3. normal weight to overweight (BMI: 18.5-29.9 kg/m2)
4. no metabolic, psychological, or neurological diseases/conditions
5. weight stable (no weight loss/gain within the past 6 mo)
6. not currently on a weight loss or other special diet (in the past 6 mo)
7. not a vegetarian
8. not pregnant
9. non-smoker

Exclusion Criteria:

1. Unhealthy
2. ages <18 or >35 years old
3. underweight or obese (BMI: <18.5 or >29.9 kg/m2)
4. metabolic, psychological, or neurological diseases/conditions
5. not weight stable (weight loss/gain within the past 6 mo)
6. Currently on a weight loss or other special diet (in the past 6 mo)
7. A vegetarian; 8) pregnant; and 9) smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Perceived Hunger | 2 months
  During each testing day, computerized questionnaires assessing hunger will be completed prior to consuming the study breakfast beverages and every half hour afterwards until leaving the testing facility. The questions are worded as "how strong is your feeling of" with anchors of "not at all" to "extremely." Each questionnaire takes approximately 30 seconds to complete. There are 10 questionnaires per testing day. Each questionnaire was completed on a netbook computer as well as through an app on an ipod touch.
Perceived Fullness | 2 months
  During each testing day, computerized questionnaires assessing fullness will be completed prior to consuming the study breakfast beverages and every half hour afterwards until leaving the testing facility. The questions are worded as "how strong is your feeling of" with anchors of "not at all" to "extremely." Each questionnaire takes approximately 30 seconds to complete. There are 10 questionnaires per testing day. Each questionnaire was completed on a netbook computer as well as through an app on an ipod touch.
Perceived Desire to Eat | 2 months
  During each testing day, computerized questionnaires assessing desire to eat will be completed prior to consuming the study breakfast beverages and every half hour afterwards until leaving the testing facility. The questions are worded as "how strong is your feeling of" with anchors of "not at all" to "extremely." Each questionnaire takes approximately 30 seconds to complete. There are 10 questionnaires per testing day. Each questionnaire was completed on a netbook computer as well as through an app on an ipod touch.
Perceived Prospective Food Consumption | 2 months
  During each testing day, computerized questionnaires assessing how much food he/she can consume will be completed prior to consuming the study breakfast beverages and every half hour afterwards until leaving the testing facility. The questions are worded as "how strong is your feeling of" with anchors of "not at all" to "an extreme amount." Each questionnaire takes approximately 30 seconds to complete. There are 10 questionnaires per testing day. Each questionnaire was completed on a netbook computer as well as through an app on an ipod touch.
Subsequent Meal Energy Intake | 2 months
  During each testing day, 4 h after the protein shake, the participants received an ad libitum pasta lunch. They were asked to consume this within 30 min until feeling 'comfortably full.' Energy and macronutrient content will be determined.

SECONDARY OUTCOMES:
Daily Food Intake | 2 months
  The day following each testing day, a dietary recall was completed to determine daily energy and macronutrient content.

IPD SHARING:
Plan to Share IPD: No